CLINICAL TRIAL: NCT00668551
Title: Pilot Randomized Controlled Trial of Telemedicine for Individuals With Parkinson Disease in a Rural Population
Acronym: Tele-PD
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Presbyterian Homes & Services (Other)
Responsible Party: E. Ray Dorsey, MD, MBA, University of Rochester
Other Study IDs: RSRB00022923
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2009-04-13 (Estimated); Status verified 2009-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Telemedicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Telemedicine care
- 2: Standard of care

SUMMARY:
To eliminate barriers (such as travel and cost) to specialized Parkinson disease (PD) care, two movement disorder specialists at the University of Rochester will be providing telemedicine visits for patients with PD who reside in the Presbyterian Home for Central New York in New Hartford, NY, or for individuals who participate in the local support group that meets at the nursing home. Participants will attend 3 telemedicine visits at the Presbyterian Home over the course of 6 months.

We hypothesize that this telemedicine model will in time improve access to care and hence the quality of life and quality of care of individuals with PD.

DETAILED DESCRIPTION:
Study participants are recruited from the Presbyterian Home and from the Central New York Parkinson Support Group. Anyone interested will attend a screening and baseline visit at the Presbyterian Home, where they will receive baseline surveys and a motor assessment. Eligible participants will be randomized to receive either telemedicine or standard of care.

Each telemedicine visit (Month 1, Month 3, Month 6) will take place in a 1:1 fashion between the study participant and the physician investigator - one of two movement disorder specialists from the University of Rochester - via televideo linkage, and will last approximately 30-60 minutes. The study participant will be observed by the physician investigator and she/he will be accompanied by a Presbyterian Home staff member to ensure safety throughout the telemedicine visit. The visit will be structured much the same as a standard clinical visit and will include:

* Study participant's update on his or her clinical condition
* Review of current medications, which will be provided in advance of the visit
* Review and update of medical and social histories
* Vital signs, including weight (provided by the Presbyterian Home staff)
* Pertinent neurological exam, including a modified motor examination led by physician investigator
* Assessment of current clinical state
* Dictated recommendations including a letter to the attending physician for ongoing clinical care, including changes to the PD medications

Participants assigned to the control group will receive their care as routinely scheduled with their own primary care physician and/or neurologist.

Staff members from the University of Rochester will return to the Presbyterian Home within one month of the six month study to complete final assessments with all study participants. These will include:

* Reportable events form
* Health care events form
* Quality of life and healthcare evaluation surveys
* Continuation of care survey
* 1:1 interviews
* Telemedicine focus groups

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age 30 years old or older
* Clinical diagnosis of idiopathic Parkinson's disease as determined by having two of the four cardinal features of PD (rest tremor, bradykinesia, cogwheel rigidity, and gait instability) and no better alternative explanation for the etiology of the symptoms
* Able to converse in English
* Willing and able to complete study requirements

Exclusion Criteria:

* Any neurological, medical, or psychiatric condition that would preclude the patient having the ability to provide informed consent or to participate in the telemedicine visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the Presbyterian Home Parkinson disease nursing home, assisted living, independent living, and adult day care populations, as well as the local PD support group that meets monthly at the Presbyterian Home.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The feasibility of telemedicine, based on participant ability to complete 75% or more of the trial visits. | 6 months

SECONDARY OUTCOMES:
Parkinson's Disease Questionnaire-39 (PDQ-39) | 6 months
EuroQol (EQ-5D) | 6 months
Geriatric Depression Scale Short Form (GDS-15) | 6 months
Modified Group Health Association of America's Consumer Satisfaction Survey (GHAA) | 6 months
Qualitative assessment, including a telemedicine focus group and 1:1 interviews with study participants | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: E. Ray Dorsey, MD, MBA, Principal Investigator — University of Rochester; Kevin Biglan, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Presbyterian Home for Central New York, Inc., New Hartford, New York, United States

REFERENCES:
- [Background] Hubble JP, Pahwa R, Michalek DK, Thomas C, Koller WC. Interactive video conferencing: a means of providing interim care to Parkinson's disease patients. Mov Disord. 1993 Jul;8(3):380-2. doi: 10.1002/mds.870080326. PMID 8341308
- [Background] Cheng EM, Swarztrauber K, Siderowf AD, Eisa MS, Lee M, Vassar S, Jacob E, Vickrey BG. Association of specialist involvement and quality of care for Parkinson's disease. Mov Disord. 2007 Mar 15;22(4):515-22. doi: 10.1002/mds.21311. PMID 17260340
- [Background] McConnochie KM, Wood NE, Kitzman HJ, Herendeen NE, Roy J, Roghmann KJ. Telemedicine reduces absence resulting from illness in urban child care: evaluation of an innovation. Pediatrics. 2005 May;115(5):1273-82. doi: 10.1542/peds.2004-0335. PMID 15867035
- [Background] Samii A, Ryan-Dykes P, Tsukuda RA, Zink C, Franks R, Nichol WP. Telemedicine for delivery of health care in Parkinson's disease. J Telemed Telecare. 2006;12(1):16-8. doi: 10.1258/135763306775321371. PMID 16438773